CLINICAL TRIAL: NCT06633328
Title: Clinical Study on the Safety and Efficacy of Donor Derived CD7 CAR-T Cell Bridging Allogeneic Hematopoietic Stem Cell Transplantation for the for Patients With Severe Aplastic Anemia
Brief Title: CD7 CAR-T Bridging to alloHSCT for Severe Aplastic Anemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2024009
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-08

CONDITIONS: Aplastic Anemia
Keywords: allo-HSCT; CD7 CAR-T
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Aplastic Anemia
  Interventions: Drug: CD7 CAR-T cells injection; Other: Allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: CD7 CAR-T cells injection — CD7 CAR T cells treat patients with severe aplastic anemia
Other: Allogeneic hematopoietic stem cell transplantation — In this study, Allogeneic hematopoietic stem cell transplantation is used as a bridge therapy to CD7 CAR T cells infusion to treat patients with severe aplastic anemia

SUMMARY:
This is a single-arm, open-label, single-center, phase I study. The primary objective is to evaluate the safety of CD7 CAR-T Bridging to allo-HSCT therapy for patients with severe aplastic anemia

DETAILED DESCRIPTION:
This is a prospective, open-label, single-center clinical trial. This study will evaluate the safety and efficacy of CD7 CAR-T Bridging to allo-HSCT in the treatment of severe aplastic anemia.The primary endpoints are dose limiting toxicity (DLT) and the incidence of treatment emergent adverse event (TEAE).

ELIGIBILITY:
Inclusion Criteria:

* Chinese expert consensus on the diagnosis and treatment of aplastic anemia（2017）, Diagnosis of severe aplastic anemia ，1. The degree of bone marrow cell proliferation < 25%, or 25%-50% but residual hematopoietic cells < 30%；2. With pancytopenia (at least two of the following peripheral blood parameters) : (1) absolute neutrophil <0.5×10^9/L; (2) Platelet count< 20×10^9/L; (3) The absolute value of reticulocytes <20×109/L;
* Suitable donors (relatives) with allogeneic HSCT indications and at least haploid allogeneic transplantation;
* Patients who are not suitable or unwilling to undergo traditional allogeneic hematopoietic stem cell transplantation;
* creatinine clearance > 60ml/min; without liver invasion, serum total bilirubin ≤ 1.5 times the upper limit of normal, and serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were both ≤ 3 times the upper limit of the normal range. If there is liver invasion, serum erythrambirubin ≤ 3 times the upper limit of normal, and serum ALT and AST are both ≤ 5 times the upper limit of the normal range;
* Echocardiogram shows left ventricular ejection fraction (LVEF) ≥ 50%;
* No active infection in the lungs, blood oxygen saturation in indoor air is ≥ 92%;
* Estimated survival time ≥ 3 months;
* ECOG performance status 0 to 1;
* Females and males of childbearing potential must agree to use adequate contraception prior to study entry, during study participation, and for 6 months after infusion (the safety of this therapy for unborn children is not known and has unknown risks);
* Those who voluntarily participated in this trial and provided informed consent;

Exclusion Criteria:

* Allergy to pre-treatment measures；
* Those with acute graft versus host disease (GvHD) or moderate to severe chronic GvHD within 4 weeks before screening; Those who have received systemic drug therapy for GvHD within 4 weeks before the reinfusion；
* History of epilepsy or other central nervous system disorders；
* Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
* Less than 100 days after allogeneic hematopoietic stem cell transplantation；
* Patients with HIV infection，Active infection of hepatitis B virus or hepatitis C virus，Uncured active infection；
* The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* Received anti-cancer chemotherapy or other drug treatment within 2 weeks prior to screening;
* Any condition that, in the opinion of the investigator, may increase the risk to the subject or interfere with the results of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2027-10-20 (Estimated); Study Completion 2027-10-20 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 days after Treatment
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Allogeneic hematopoietic stem cell transplant implantation rate | Up to 100 days after Treatment
  The proportion of the number of patients who achieved hematopoietic reconstitution to the total number of allogeneic hematopoietic stem cell transplantation patients in the same period.
Time to neutrophil and platelet engraftment | Up to 30 days after Treatment
  The time for neutrophils and platelets to reach the implantation criteria after stem cell reinfusion
Disease-feesurvival，DFS | Up to 2 years after Treatment
  The proportion of disease-free patients who survived to the total number of patients who transplanted allogeneic hematopoietic stem cells during the same period.
Overall survival, OS | Up to 2 years after Treatment
  After transplantation until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hanzhou, Zhejiang, China